CLINICAL TRIAL: NCT05580510
Title: "An Open-label Clinical Trial to Evaluate the Safety and Efficacy of Empagliflozin and Sacubitril/Valsartan in Adult Patients With Chronic Heart Failure With Reduced Ejection Fraction Associated With Congenital Heart Disease"
Brief Title: " Evaluation of Safety and Efficacy of Empagliflozin and Sacubitril/Valsartan for CHF With Reduced Ejection Fraction in ACHD "
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-1333
Record Dates: First submitted 2022-10-04; First posted 2022-10-14 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Congenital Heart Disease; Heart Failure; Heart Failure With Reduced Ejection Fraction
Keywords: Adult congenital heart disease; Heart Failure with Reduced Ejection Fraction; Empagliflozin; Sacubitril-valsartan
MeSH Terms: conditions — Heart Defects, Congenital; Heart Failure | interventions — sacubitril; Valsartan; sacubitril and valsartan sodium hydrate drug combination; BID protein, human; empagliflozin

STUDY DESIGN:
Intervention Model Description: Open-label randomized clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Conventional treatment of Heart failure and Sacubitril/Valsartan (Active Comparator): Patients will receive conventional treatment consisting of spironolactone 25 mg orally every 24 hours (maximum dose 50 mg every 24 hours) or eplerenone 25 mg orally every 24 hours (maximum dose 50 mg every 24 hours); beta-blockers: bisoprolol 1.5 mg orally every 24 hours (maximum dose 10 mg every 24 hours) or metoprolol succinate 12.5 mg every 24 hours orally (maximum dose 200 mg every 24 hours) or carvedilol 3125 mg every 24 hours (maximum dose 25 mg every 24 hours) or ivabradine 5 mg every 12 hours (maximum dose 7.5 mg every 12 hours); diuretics: furosemide 20 to 400 mg orally every 24 hours or bumetanide 1 to 15 mg orally every 24 hours and/or chlorthalidone 25 mg orally every 24 hours.
  Additionally, patients will receive Sacubitril/Valsartan, with the intention to titrate up to 49 mg/51 mg orally every 12 hours.
  Interventions: Drug: Sacubitril 49 MG / Valsartan 51 MG [Entresto] BID
- Conventional treatment plus Empagliflozin and Sacubitril/valsartan (Experimental): Patients will receive conventional treatment consisting of spironolactone 25 mg orally every 24 hours (maximum dose 50 mg every 24 hours) or eplerenone 25 mg orally every 24 hours (maximum dose 50 mg every 24 hours); beta-blockers: bisoprolol 1.5 mg orally every 24 hours (maximum dose 10 mg every 24 hours) or metoprolol succinate 12.5 mg every 24 hours orally (maximum dose 200 mg every 24 hours) or carvedilol 3125 mg every 24 hours (maximum dose 25 mg every 24 hours) or ivabradine 5 mg every 12 hours (maximum dose 7.5 mg every 12 hours); diuretics: furosemide 20 to 400 mg orally every 24 hours or bumetanide 1 to 15 mg orally every 24 hours and/or chlorthalidone 25 mg orally every 24 hours.
  Additionally, patients will use Sacubitril/Valsartan, with the intention to titrate up to 49 mg/51 mg orally every 12 hours and Empagliflozin 10 mg orally every 24 hours.
  Interventions: Drug: Sacubitril 49 MG / Valsartan 51 MG [Entresto] BID; Drug: Empagliflozin 10 MG OD
- Conventional treatment plus Empagliflozin (Experimental): Patients will receive conventional treatment consisting of spironolactone 25 mg orally every 24 hours (maximum dose 50 mg every 24 hours) or eplerenone 25 mg orally every 24 hours (maximum dose 50 mg every 24 hours); beta-blockers: bisoprolol 1.5 mg orally every 24 hours (maximum dose 10 mg every 24 hours) or metoprolol succinate 12.5 mg every 24 hours orally (maximum dose 200 mg every 24 hours) or carvedilol 3125 mg every 24 hours (maximum dose 25 mg every 24 hours) or ivabradine 5 mg every 12 hours (maximum dose 7.5 mg every 12 hours); diuretics: furosemide 20 to 400 mg orally every 24 hours or bumetanide 1 to 15 mg orally every 24 hours and/or chlorthalidone 25 mg orally every 24 hours.
  Additionally, patients will use Empagliflozin 10 mg orally every 24 hours.
  Interventions: Drug: Empagliflozin 10 MG OD

INTERVENTIONS:
Drug: Sacubitril 49 MG / Valsartan 51 MG [Entresto] BID — This group of patients will receive the conventional treatment of heart failure according to the "2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure" and Sacubitril/Valsartan as an active comparator.
  Other Names: Entresto
  Arms: Conventional treatment of Heart failure and Sacubitril/Valsartan; Conventional treatment plus Empagliflozin and Sacubitril/valsartan
Drug: Empagliflozin 10 MG OD — This group of patients will receive the conventional treatment of heart failure according to the "2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure" and Empagliflozin as an experimental drug.
  Other Names: Jardiance
  Arms: Conventional treatment plus Empagliflozin; Conventional treatment plus Empagliflozin and Sacubitril/valsartan

SUMMARY:
The treatment of adult patients with congenital heart disease (ACHD) and heart failure (HF) represents a great challenge since, to date, there is no standardized guideline for this specific population. Although new treatments for HF have been proposed, such as Sodium-glucose Cotransporter-2 (SGLT2) Inhibitors and neprilisin and angiotensin receptor inhibitors, the benefit of these drugs in patients with HF associated with congenital heart disease in adults has not yet been demonstrated. For this reason, this study pretends to evaluate the efficacy of empagliflozin and sacubitril/valsartan in this population.

DETAILED DESCRIPTION:
A 12-week randomized, open label, active-controlled trial to explore the effects of once-daily empagliflozin 10 mg and/or sacutril/valsartan 49 mg/51 mg in the reduction of systemic ventricular volumes (end-diastolic and end-systolic) in adult patients with HF associated with congenital heart disease.

ELIGIBILITY:
Inclusion Criteria:

* NYHA functional class II-IV
* Diagnosis of CHD: repaired, palliated or without previous treatment
* Systemic ventricular ejection fraction <40%
* Without unplanned hospital admissions within 3 months prior to randomization
* The participant is willing and able to give informed consent for participation in the study

Exclusion Criteria:

* Pregnant and postpartum women
* Breastfeeding women during the study
* History of drug allergy to any SGLT-2 inhibitor and/or sacubitril/valsartan
* Previous administration of a drug regimen including an SGLT-2 inhibitor and/or sacubitril/valsartan
* Intellectual or physical disability that impedes the subject to perform the 6 minute walk-test
* Patients with any contraindication to SGLT-2 inhibitor and/or sacubitril/valsartan
* Medical history of myocardial infarction, cardiac surgery or fulminant myocarditis within the last three months
* Medical history of type 1 diabetes mellitus
* Medical history of hypertensive crisis in the previous 6-months
* Medical history of cardiogenic shock or heart failure decompensation in the previous 6-months
* Medical history of heart transplantation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-02-06 (Estimated); Primary Completion 2023-07-28 (Estimated); Study Completion 2024-03-29 (Estimated)

PRIMARY OUTCOMES:
3D echocardiographic systemic ventricular end-diastolic volume index | Twelve weeks
  Change of 8.2 ml or greater in systemic ventricular end-diastolic volume index measured by 3D echocardiogram.
3D echocardiographic systemic ventricular end-systolic volume index | Twelve weeks
  Change of 6.0 ml or greater in end-systolic volume index measured by 3D echocardiogram.

SECONDARY OUTCOMES:
Functional class | Twelve weeks
  A clinically relevant change of greater than or equal to 5 points from baseline score in the functional class measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ). This questionnaire evaluates 23 elements and is divided into 7 different domains. The score will interpreted as follows:
  0-24 points: very poor to poor 25-49 points: poor to fair 50-74 points: fair to good 75-100 points: good to excellent
Pulmonary congestion | Twelve weeks
  Change in pulmonary B score measured by the quantification and characteristics of B-lines seen with pulmonary ultrasound assessing 8 regions total using the following scoring system:
  0 points: less than 3 B-lines per zone
  1 point: greater than or equal to 3 B-lines per zone
6-minute walking test | Twelve weeks
  Difference in meters walked in the 6-minute walking test.
Echocardiographic ejection fraction from the systemic ventricle | Twelve weeks
  A change in the percentage of ejection fraction from the systemic ventricle measured by echocardiogram.
Echocardiographic longitudinal overall strain | Twelve weeks
  A change in the percentage of longitudinal overall strain measured by echocardiogram at baseline and after treatment.
NT-proBNP | Twelve weeks
  Change in NT-proBNP values.
Systemic venous congestion | Twelve weeks
  Change in VExUS grading system measured by the diameter of the inferior vena cava in cm and Doppler pattern abnormalities on hepatic, portal and intra-renal veins using the following scoring system:
  No congestion (0): IVC less than 2 cm Mild (1): IVC greater than or equal to 2cm and any normal or mildly abnormal patterns Moderate (2): IVC greater than or equal to 2cm and ONE severely abnormal pattern Severe (3): IVC greater than or equal to 2 cm and more than or equal to TWO severely abnormal patterns

CONTACTS AND LOCATIONS:
Overall Officials: Edgar Garcia-Cruz, MD, Principal Investigator — National Institute of Cardiology Ignacio Chavez; Montserrat Villalobos-Pedroza, MD, Study Chair — National Institute of Cardiology Ignacio Chavez; Gian Jimenez-Rodriguez, MD, Study Chair — National Institute of Cardiology Ignacio Chávez; Carlos Guizar-Sanchez, MD, Study Director — National Institute of Cardiology Ignacio Chávez
Locations (1):
- National Institute of Cardiology Ignacio Chavez, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Velazquez EJ, Morrow DA, DeVore AD, Duffy CI, Ambrosy AP, McCague K, Rocha R, Braunwald E; PIONEER-HF Investigators. Angiotensin-Neprilysin Inhibition in Acute Decompensated Heart Failure. N Engl J Med. 2019 Feb 7;380(6):539-548. doi: 10.1056/NEJMoa1812851. Epub 2018 Nov 11. PMID 30415601
- [Background] Hu J, Wu Y, Zhou X, Wang X, Jiang W, Huo J, Shan Q. Beneficial Effects of Sacubitril/Valsartan at Low Doses in an Asian Real-World Heart Failure Population. J Cardiovasc Pharmacol. 2020 Oct;76(4):445-451. doi: 10.1097/FJC.0000000000000873. PMID 33030857
- [Background] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2021 Sep 21;42(36):3599-3726. doi: 10.1093/eurheartj/ehab368. No abstract available. PMID 34447992
- [Background] Budts W, Roos-Hesselink J, Radle-Hurst T, Eicken A, McDonagh TA, Lambrinou E, Crespo-Leiro MG, Walker F, Frogoudaki AA. Treatment of heart failure in adult congenital heart disease: a position paper of the Working Group of Grown-Up Congenital Heart Disease and the Heart Failure Association of the European Society of Cardiology. Eur Heart J. 2016 May 7;37(18):1419-27. doi: 10.1093/eurheartj/ehv741. Epub 2016 Jan 18. No abstract available. PMID 26787434
- [Background] Marelli, A. Gatzoulis, M. Gary, D. Webb, Piers E.F. Daubeney. Adults With Congenital Heart Disease: A Growing Population. Chapter 1 Part I General Principles. Diagnosis and Management of Adult Congenital Heart Disease. (2017): 2-9.
- [Background] Stout KK, Broberg CS, Book WM, Cecchin F, Chen JM, Dimopoulos K, Everitt MD, Gatzoulis M, Harris L, Hsu DT, Kuvin JT, Law Y, Martin CM, Murphy AM, Ross HJ, Singh G, Spray TL; American Heart Association Council on Clinical Cardiology, Council on Functional Genomics and Translational Biology, and Council on Cardiovascular Radiology and Imaging. Chronic Heart Failure in Congenital Heart Disease: A Scientific Statement From the American Heart Association. Circulation. 2016 Feb 23;133(8):770-801. doi: 10.1161/CIR.0000000000000352. Epub 2016 Jan 19. No abstract available. PMID 26787728
- [Background] Konstatinos D. Alonso- González R, D'alto M. Heart Failure, Exercise Intolerance and Physical Training. Chapter 7, Part I General Principles. Diagnosis and Management of Adult Congenital Heart Disease. (2017): 77-87.
- [Background] Arnaert S, De Meester P, Troost E, Droogne W, Van Aelst L, Van Cleemput J, Voros G, Gewillig M, Cools B, Moons P, Rega F, Meyns B, Zhang Z, Budts W, Van De Bruaene A. Heart failure related to adult congenital heart disease: prevalence, outcome and risk factors. ESC Heart Fail. 2021 Aug;8(4):2940-2950. doi: 10.1002/ehf2.13378. Epub 2021 May 7. PMID 33960724
- [Result] Jhund PS, Ponikowski P, Docherty KF, Gasparyan SB, Bohm M, Chiang CE, Desai AS, Howlett J, Kitakaze M, Petrie MC, Verma S, Bengtsson O, Langkilde AM, Sjostrand M, Inzucchi SE, Kober L, Kosiborod MN, Martinez FA, Sabatine MS, Solomon SD, McMurray JJV. Dapagliflozin and Recurrent Heart Failure Hospitalizations in Heart Failure With Reduced Ejection Fraction: An Analysis of DAPA-HF. Circulation. 2021 May 18;143(20):1962-1972. doi: 10.1161/CIRCULATIONAHA.121.053659. Epub 2021 Apr 9. PMID 33832352
- [Result] Packer M, Anker SD, Butler J, Filippatos G, Pocock SJ, Carson P, Januzzi J, Verma S, Tsutsui H, Brueckmann M, Jamal W, Kimura K, Schnee J, Zeller C, Cotton D, Bocchi E, Bohm M, Choi DJ, Chopra V, Chuquiure E, Giannetti N, Janssens S, Zhang J, Gonzalez Juanatey JR, Kaul S, Brunner-La Rocca HP, Merkely B, Nicholls SJ, Perrone S, Pina I, Ponikowski P, Sattar N, Senni M, Seronde MF, Spinar J, Squire I, Taddei S, Wanner C, Zannad F; EMPEROR-Reduced Trial Investigators. Cardiovascular and Renal Outcomes with Empagliflozin in Heart Failure. N Engl J Med. 2020 Oct 8;383(15):1413-1424. doi: 10.1056/NEJMoa2022190. Epub 2020 Aug 28. PMID 32865377
- [Result] Bauersachs J. Heart failure drug treatment: the fantastic four. Eur Heart J. 2021 Feb 11;42(6):681-683. doi: 10.1093/eurheartj/ehaa1012. No abstract available. PMID 33447845
- [Result] Lee MMY, Brooksbank KJM, Wetherall K, Mangion K, Roditi G, Campbell RT, Berry C, Chong V, Coyle L, Docherty KF, Dreisbach JG, Labinjoh C, Lang NN, Lennie V, McConnachie A, Murphy CL, Petrie CJ, Petrie JR, Speirits IA, Sourbron S, Welsh P, Woodward R, Radjenovic A, Mark PB, McMurray JJV, Jhund PS, Petrie MC, Sattar N. Effect of Empagliflozin on Left Ventricular Volumes in Patients With Type 2 Diabetes, or Prediabetes, and Heart Failure With Reduced Ejection Fraction (SUGAR-DM-HF). Circulation. 2021 Feb 9;143(6):516-525. doi: 10.1161/CIRCULATIONAHA.120.052186. Epub 2020 Nov 13. PMID 33186500
- [Result] Nougue H, Pezel T, Picard F, Sadoune M, Arrigo M, Beauvais F, Launay JM, Cohen-Solal A, Vodovar N, Logeart D. Effects of sacubitril/valsartan on neprilysin targets and the metabolism of natriuretic peptides in chronic heart failure: a mechanistic clinical study. Eur J Heart Fail. 2019 May;21(5):598-605. doi: 10.1002/ejhf.1342. Epub 2018 Dec 6. PMID 30520545